CLINICAL TRIAL: NCT03454295
Title: Improving Palliative Care of Caregivers of Patients With Glioblastoma
Brief Title: Easing Psychosocial Burden for Informal Caregivers
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 18-075
Record Dates: First submitted 2018-02-14; First posted 2018-03-05 (Actual); Last update posted 2024-04-01 (Actual); Status verified 2024-03

CONDITIONS: Glioblastoma
Keywords: Cancer Caregivers; Caregiver; Caregivers; Memorial Sloan Kettering Cancer Center; 18-075
MeSH Terms: conditions — Glioblastoma | interventions — Focus Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Part I (Experimental): Focus group (Part 1) of four to ten GBM ICs bereaved at least one year to help determine our recruitment strategy. Participants will be asked to reflect on their caregiving experience and specifically, when the receipt of a supportive intervention that addresses existential distress would have been most appropriate and well received. Should consensus among participants be reached (e.g., if the majority report that being approached at time of their loved one's cancer recurrence would have been the optimal time for enrollment), we will target our enrollment timeline to this point (and this timeline will be reflected in amended inclusion criteria). If no consensus is reached, the study staff will enroll ICs at all points in the caregiving trajectory and revisit the appropriateness of various points of contact during the Part 2 individual interviews.
  Interventions: Behavioral: Focus Group
- Part II (Experimental): In Part 2, we will recruit 60 ICs of patients with GBM who will be randomized to receive either MCP-C or EUC. MCP-C will be delivered individually over 7 1-hour-long sessions within 7 - 14 weeks.
  Interventions: Behavioral: Meaning-Centered Psychotherapy for Cancer Caregivers / MCP-C; Behavioral: Enhanced Usual Care / EUC

INTERVENTIONS:
Behavioral: Focus Group — Participants will be asked to reflect on their caregiving experience and specifically, when the receipt of a supportive intervention that addresses existential distress would have been most appropriate and well received.
  Arms: Part I
Behavioral: Meaning-Centered Psychotherapy for Cancer Caregivers / MCP-C — MCP-C is structured as a 7-session (1-hour weekly or biweekly sessions) individual intervention that utilizes a mixture of didactics, discussion and experiential exercises that focus around particular themes related to meaning and cancer caregiving
  Arms: Part II
Behavioral: Enhanced Usual Care / EUC — The "enhancement" to usual care in this study involves the inclusion of screening and targeted referral components as suggested by Reynolds et al. [79]. Research study assistants conducting the screening and providing feedback and referrals will be trained in the NCCN guidelines for distress management and will discuss the screening results and associated recommendations with the study PI (NCCN) [63]. As of November, 2017, ICs of patients seen in the Neurology Service at MSKCC are not consistently screened for distress and offered targeted referrals. Participants randomized to EUC will receive feedback about their level of distress (based on the Distress Thermometer administered at screening) after randomization. Within a week of randomization, and post-baseline, the study RSA will send EUC participants appropriate targeted referrals based on levels of distress and problem areas endorsed.
  Arms: Part II

SUMMARY:
The overall goal of this study is to determine the best time to offer Meaning-Centered Psychotherapy (MCP), an intervention that has proven to be helpful in improving spiritual well-being and decreasing existential distress among patients with advanced cancer, to caregivers. (MCP has also been shown to be an appropriate method of attending to the palliative or comfort care needs of caregivers of patients with cancer. Studies show that the psychological burden associated with caring for a patient with advanced cancer is often greater than that experienced by the patients themselves.) The investigators would also like to find out about caregivers initial impressions of MCP-C, Meaning-Centered Psychotherapy for Cancer Caregivers, so that the intervention can be adjusted to meet the unique needs of caregivers of patients with Glioblastoma.

ELIGIBILITY:
Inclusion Criteria:

Part I Focus group GBM informal caregivers (ICs):

* English-speaking as English proficiency screener and in the best judgment of the consenting professional. This is due to the focus groups being managed in English and the use of certain validated questionnaires only being available in English.
* Age > 18
* IC to an MSKCC patient with GBM who died a year or more ago

Part II Randomized Intervention of GBM ICs:

* English-speaking as per English proficiency screener and in the best judgment of the consenting professional
* Current ICs to a patient with GBM
* Age ≥ 18
* Score of > 4 on the Distress Thermometer (DT) and indication that this distress is related in some way to the caregiving role per self-report

Exclusion Criteria:

* In the judgment of the consenting professional, clinician or PI and/or as per medical record, severe psychopathology or cognitive impairment likely to interfere with the participation or completion of the protocol or ability to provide meaningful information
* Another family member of caregiver to the same patients is currently enrolled in the study
* Ultimately, if interested, all caregivers who decline participation or are ineligible for the study for any reason, including because another caregiver of the patient is currently enrolled in the study, will be offered referrals to the MSKCC Counseling Center and to local mental health providers

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2018-02-12 (Actual); Primary Completion 2024-03-26 (Actual); Study Completion 2024-03-26 (Actual)

PRIMARY OUTCOMES:
Feasibility of Meaning-Centered Psychotherapy for Cancer Caregivers (MCP-C) delivered to caregivers of participants with GBM | 1 year
  Feasibility will be measured by our ability to recruit our target sample of 60 ICs within the 1-year enrollment period. Our feasibility target for completion of follow-up assessments if 80% at T2 and 60% at T3, based on typical assessment completion rates in other psychosocial intervention studies conducted at our institution.
Acceptability of Meaning-Centered Psychotherapy for Cancer Caregivers (MCP-C) delivered to caregivers of participants with GBM | 1 year
  Acceptability will be informed by the MCP-C completion rate and Phase 2 semi-structured interviews (deemed acceptable if at least 40% complete all psychotherapy sessions).

CONTACTS AND LOCATIONS:
Overall Officials: Allison Applebaum, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (3):
- United States (3):
  - Memorial Sloan Kettering Commack (Consent only), Commack, New York
  - Memorial Sloan Kettering Westchester (Consent only), Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://mskcc.org